CLINICAL TRIAL: NCT02435329
Title: Bone Metabolism and Endothelial Function in Patients With Type 2 Diabetes Mellitus and Charcot Foot - an Observational Comparative Study
Brief Title: Microcirculation and Bone Metabolism in Patients With Type 2 Diabetes Mellitus and Charcot Foot - A Pilot Study
Status: Completed | Type: Observational
Sponsor: Tameside General Hospital (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: Charcodiab13; 15/NI/0043 (Other: HSC REC A)
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Angiopathies; Bone Diseases, Metabolic
MeSH Terms: conditions — Diabetic Angiopathies; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Analysis of serum samples for markers of endothelial function, inflammation and bone metabolism
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy volunteers: 10 healthy volunteers
  * Anthropometric measures: Height, weight, BMI, waist circumference
  * Vital parameters: supine and standing blood pressure, pulse, respiratory rate and temperature
  * Laboratory assessment that includes markers of endothelial activation, inflammation and bone metabolism.
  * Assessment of skin microcirculation with Laser Doppler Iontophoresis
  * Assessment of calcaneal bone mineral density (BMD) with Bone Sonometer (ultrasound)
  * Advanced glycation end-products will be assessed by an AGE reader which uses the technique of skin autofluorescence
  Interventions: Other: Baseline comparison of microcirculation and bone metabolism
- Type 2 diabetes without neuropathy: 10 patients
  * Anthropometric measures: Height, weight, BMI, waist circumference
  * Vital parameters: supine and standing blood pressure, pulse, respiratory rate and temperature
  * Laboratory assessment that includes markers of endothelial activation, inflammation and bone metabolism.
  * Assessment of skin microcirculation with Laser Doppler Iontophoresis
  * Assessment of calcaneal bone mineral density (BMD) with Bone Sonometer (ultrasound)
  * Advanced glycation end-products will be assessed by an AGE reader which uses the technique of skin autofluorescence
  Interventions: Other: Baseline comparison of microcirculation and bone metabolism
- Type 2 diabetes with painful neuropathy: 10 patients
  * Anthropometric measures: Height, weight, BMI, waist circumference
  * Vital parameters: supine and standing blood pressure, pulse, respiratory rate and temperature
  * Laboratory assessment that includes markers of endothelial activation, inflammation and bone metabolism.
  * Assessment of skin microcirculation with Laser Doppler Iontophoresis
  * Assessment of calcaneal bone mineral density (BMD) with Bone Sonometer (ultrasound)
  * Advanced glycation end-products will be assessed by an AGE reader which uses the technique of skin autofluorescence
  Interventions: Other: Baseline comparison of microcirculation and bone metabolism
- Type 2 diabetes with painless neuropathy: 10 patients
  * Anthropometric measures: Height, weight, BMI, waist circumference
  * Vital parameters: supine and standing blood pressure, pulse, respiratory rate and temperature
  * Laboratory assessment that includes markers of endothelial activation, inflammation and bone metabolism.
  * Assessment of skin microcirculation with Laser Doppler Iontophoresis
  * Assessment of calcaneal bone mineral density (BMD) with Bone Sonometer (ultrasound)
  * Advanced glycation end-products will be assessed by an AGE reader which uses the technique of skin autofluorescence
  Interventions: Other: Baseline comparison of microcirculation and bone metabolism
- Type 2 diabetes with Charcot foot: 10 patients
  * Anthropometric measures: Height, weight, BMI, waist circumference
  * Vital parameters: supine and standing blood pressure, pulse, respiratory rate and temperature
  * Laboratory assessment that includes markers of endothelial activation, inflammation and bone metabolism.
  * Assessment of skin microcirculation with Laser Doppler Iontophoresis
  * Assessment of calcaneal bone mineral density (BMD) with Bone Sonometer (ultrasound)
  * Advanced glycation end-products will be assessed by an AGE reader which uses the technique of skin autofluorescence
  Interventions: Other: Baseline comparison of microcirculation and bone metabolism

INTERVENTIONS:
Other: Baseline comparison of microcirculation and bone metabolism — Baseline comparison of microcirculation and bone metabolism among the 5 different groups

SUMMARY:
This study is part of a research project for a University MD Program. This is an observational study aimed at comparing the differences in bone metabolism and microcirculation in patients with type 2 diabetes mellitus (with and without diabetic neuropathy and Charcot foot) with healthy subjects.

Diabetes is gradually becoming a global epidemic along with its associated complications. Diabetes can affect several systems in our body particularly the eyes, nerves and the kidneys. The damaging effects occur at the level of the small blood vessels (microcirculation) that supply these vital structures. Normally, the inner lining of these blood vessels (endothelium) plays a very important role in maintaining adequate blood flow. The endothelium releases a chemical substance called nitric oxide, which relaxes these small blood vessels thereby ensuring sufficient blood supply to these key structures. Nitric oxide also prevents blockage of these vessels. Any form of metabolic stress like hyperglycaemia (raised blood sugar as seen in diabetes) can cause abnormal changes in the normal behaviour of the endothelium (endothelial dysfunction). Therefore hyperglycaemia promotes endothelial dysfunction by lowering nitric oxide levels, which may lead to diabetic complications like diabetic retinopathy (eye damage), nephropathy (kidney damage) or neuropathy (nerve damage).

In addition, patients with diabetes also suffer from osteoporosis (thinning of bones). Osteoporosis is a bone disorder characterised by a reduction in bone mineral content leading to an increased risk of developing fractures. The increased risk of fractures in patients with type 2 diabetes is attributed to poor bone quality resulting from the harmful effects of high blood glucose. Studies have also shown that nitric oxide has a bone protective effect as demonstrated by its ability to prevent bone fragmentation and improve bone strength.

Study of markers of endothelial function and bone metabolism will facilitate a better understanding about the origin of diabetic complications. This will aid in the development of novel therapeutic agents that target the harmful triggers in diabetes and eventually may prevent and retard the onset of the debilitating diabetic complications.

DETAILED DESCRIPTION:
This is an observational study aimed at observing and comparing differences in bone metabolism and microcirculation in patients with type 2 diabetes and healthy controls.

In this study, 50 participants will be recruited and then categorised into the following groups:

1. Control group: 10 healthy volunteers (Hospital staff and spouses/ partners of patients will volunteer as healthy subjects)
2. Type 2 diabetic patients without neuropathy: 10
3. Type 2 diabetic patients with neuropathy:

   * 10 patients with painless neuropathy
   * 10 patients with painful neuropathy
4. Type 2 diabetic patients with unilateral Charcot foot: 10

Visit Schedule The estimated time for enrollment of patients will be within 3 months. The duration of the study is 5 months.

Screening (-2 Weeks): To assess for eligibility. This will include informed consent process, medical history and physical examination, screening for neuropathy and routine bloods. Laboratory work-up done at screening will be considered for data analysis.

Visit 1 - Baseline visit

* Anthropometric measures: Height, weight, BMI, waist circumference
* Vital parameters: supine and standing blood pressure, pulse, respiratory rate and temperature
* Laboratory assessment that includes markers of endothelial activation, inflammation and bone metabolism.

  * Markers of endothelial activation will be investigated using systemic protein suspension array technology. For e.g. adhesion molecules like ICAM, VCAM and inflammatory molecules.
  * Nitric oxide will be analysed using Griess assay
  * Bone turnover markers [e.g., P1NP (Procollagen type 1 amino terminal propeptide), CTX (C-terminal cross-linked telopeptide of type-I collagen), Sclerostin, RANKL (receptor activator for nuclear factor (NF)-kB (RANK) ligand), OPG (osteoprotegerin), OPN (osteopontin), OCN (osteocalcin), BMP4 (Bone morphogenetic protein 4) and TGF-1β(Transforming growth factor-1β) - using ELISA (enzyme-linked immunosorbent assay).
  * IL-6 - Interleukin-6, an inflammatory cytokine implicated in osteoporosis (using ELISA)
* Assessment of skin microcirculation with Laser Doppler Iontophoresis
* Assessment of calcaneal bone mineral density (BMD) with Bone Sonometer (ultrasound)
* Advanced glycation end-products will be assessed by an AGE reader which uses the technique of skin autofluorescence

Clinical Procedures

Assessment of the microcirculation with Laser Doppler Iontophoresis:

A standard measurement of microcirculation is laser Doppler iontophoresis, which is used by several research institutes. In this trial the skin microcirculation will be measured on the dorsum of the foot using a Perimed Laser Doppler imager and iontophoresis system.

Endothelial-mediated vasodilation will be measured by the iontophoresis of acetylcholine, while sodium nitroprusside will be used to measure endothelium-independent vasodilation. The iontophoresis system consists of an ION chamber (iontophoresis delivery vehicle device) that sticks firmly to the skin and a reference electrode. The response in blood flow will be imaged and quantified using the Perimed Laser Doppler Imager (PeriScan PIMII; Perimed, Sweden).

Analysis of AGE:

An AGE reader, which utilizes the principle of skin autofluorescence, will measure the accumulation of AGE in the skin. This validated device provides a real-time, non-invasive assessment of cardiovascular risk for chronic diseases like Diabetes, renal failure, cardiovascular disease, etc. AGE-modified proteins have autofluorescent properties and when excited by ultraviolet (UV) light they emit fluorescence in particular wavelengths. The levels of AGE in skin correlate with AGE levels in blood.

The volar aspect of the forearm will be placed on the AGE reader, which is equipped with a UV light source. The UV light triggers AGE in skin, after penetrating 1mm of the dermis, to emit autofluorescence that is then detected by the AGE reader. The intensity of fluorescence correlates with the quantity of AGE in the skin.

Assessment of calcaneal BMD:

This is a simple and convenient method to assess peripheral BMD and assess fracture risk. The device used is a quantitative ultrasound called Sahara Clinical Bone Sonometer (Sahara Clinical Bone Sonometer; Hologic, Waltham, MA). The calcaneus is the preferred peripheral site to assess fracture risk. This device uses ultrasound waves to determine the BMD of the calcaneus. In this procedure, once the bare heel is placed in the device, the BMD is calculated within 30 seconds and the results are then generated on paper by the device.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects aged between 40-75 years

  * Healthy subjects or non-diabetic subjects for the control group.
  * A diagnosis of type 2 DM based on one of the following criteria (ADA - 2010):
* Fasting plasma glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L) or
* 2-h plasma glucose ≥ 200 mg/dl (11.1 mmol/L) during an OGTT or
* Classic symptoms of hyperglycaemia or hyperglycaemic crisis with a random plasma glucose ≥ 200 mg/dL (11.1 mmol/L).

  * Patients on treatment for type 2 diabetes mellitus
  * Presence of diabetic neuropathy will be confirmed when 2 of the following neurological tests are positive on examination (vibration perception threshold, 10 gm. monofilament, 128 Hz tuning fork, ankle reflex, pin-prick)
  * Painful diabetic neuropathy diagnosed according to LANSS (Leeds Assessment of Neuropathic Symptoms and Signs) scoring
  * For patients with chronic Charcot foot, the diagnosis should be confirmed by clinical judgment and by radiologic examination - X-ray, technetium-labeled bisphosphonate bone scan or MRI)

Exclusion Criteria:

* • At screening, age below 40 years and above 75 years.

  * Type 1 diabetes mellitus (patients with a history of ketoacidosis, age of onset of DM before 25 years of age, BMI <21 kg/m2 and use of insulin without a concomitant oral hypoglycemic agent)
  * Major cardiovascular complications within 3 months prior to screening
  * Recent history of smoking within the last 6 months
  * Scars, tattoos or rashes over the forearm
  * Recent or current oral steroid therapy or topical steroids applied to the forearm
  * Patients with uncontrolled hypertension (systolic blood pressure [SBP] > 160/90 mmHg) or hypotension (SBP ≤ 100 mm Hg or a diastolic BP of ≤60 mm Hg) at screening.
  * History of general systemic illness including cardiac, hepatic or renal insufficiency
  * Patients with renal insufficiency characterized by a creatinine clearance of less than 60 ml/min or a serum creatinine of more than 130 μmol/l
  * Receiving treatment for inflammatory disease or malignancy
  * Other non-diabetic causes of neuropathy
  * History of chronic alcohol consumption
  * History of metabolic bone disorders (Osteoporosis, Paget's disease, etc.) or treatment for bone disorders (past or current treatment for osteoporosis, bisphosphonate therapy within the last 3 years)
  * History of malignancy
  * History of active foot ulcers
  * History of concomitant therapy that may interfere with bone metabolism e.g. glucocorticoids (within the last 3 months), hormone replacement therapy (in the last 12 months), SERM (selective oestrogen receptor modulator), thiazolidinedione, anticonvulsant use
  * Receiving drugs that fluoresce (e.g., Doxorubicin, Daunomycin, Camptothecin, Protoporphyrin, Fluoroquinolones, Tetracycline, Hydroxychloroquine or Quinidine)
  * History of photosensitivity reactions (e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity
  * Simultaneous participation in other clinical trials or involvement in another research trial involving an investigational product in the past 12 weeks.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 patients with type 2 diabetes mellitus will be considered eligible for the study. Patients with a previous diagnosis of type 2 diabetes mellitus and newly diagnosed type 2 DM seen at Tameside Hospital will be recruited into the study. In addition, eligible patients will be identified and referred from University Hospital of South Manchester (UHSM) and appropriate GP practices (from Oldham, Tameside and Wythenshawe).
  Source of healthy controls: Hospital staff and spouses/ partners of patients will volunteer as healthy subjects.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Impaired endothelial function in patients with type 2 DM with/ without diabetic neuropathy and Charcot foot compared to their healthy counterparts as measured by: | At baseline
  Endothelial-dependent and independent vasodilatations
Impaired endothelial function in patients with type 2 DM with/ without diabetic neuropathy and Charcot foot compared to their healthy counterparts as measured by: | at baseline
  Markers of endothelial activation, which include adhesion molecules like ICAM, VCAM and inflammatory molecules.
Impaired endothelial function in patients with type 2 DM with/ without diabetic neuropathy and Charcot foot compared to their healthy counterparts as measured by: | at baseline
  Serum Nitric oxide
Impaired endothelial function in patients with type 2 DM with/ without diabetic neuropathy and Charcot foot compared to their healthy counterparts as measured by: | at baseline
  Advanced glycation end-products

SECONDARY OUTCOMES:
Impaired bone metabolism in patients with type 2 DM with/ without diabetic neuropathy and Charcot foot compared to their healthy counterparts as assessed by: | At baseline
  Bone turnover markers like P1NP, CTX, Sclerostin, RANKL, OPG, OPN, OCN, BMP4 and TGF-1β.
Impaired bone metabolism in patients with type 2 DM with/ without diabetic neuropathy and Charcot foot compared to their healthy counterparts as assessed by: | At baseline
  Calcaneal bone mineral density (BMD)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Jude, MD, MRCP, Principal Investigator — Tameside Hospital NHS Foundation Trust
Locations (1):
- Tameside Hospital NHS Foundation Trust, Ashton-under-Lyne, Greater Manchester, United Kingdom

REFERENCES:
- [Background] Mascarenhas JV, Jude EB. Pathogenesis and medical management of diabetic Charcot neuroarthropathy. Med Clin North Am. 2013 Sep;97(5):857-72. doi: 10.1016/j.mcna.2013.05.002. PMID 23992897
- [Background] Hofbauer LC, Brueck CC, Singh SK, Dobnig H. Osteoporosis in patients with diabetes mellitus. J Bone Miner Res. 2007 Sep;22(9):1317-28. doi: 10.1359/jbmr.070510. PMID 17501667
- [Background] Vestergaard P. Discrepancies in bone mineral density and fracture risk in patients with type 1 and type 2 diabetes--a meta-analysis. Osteoporos Int. 2007 Apr;18(4):427-44. doi: 10.1007/s00198-006-0253-4. Epub 2006 Oct 27. PMID 17068657
- [Background] Wimalawansa SJ. Nitric oxide: new evidence for novel therapeutic indications. Expert Opin Pharmacother. 2008 Aug;9(11):1935-54. doi: 10.1517/14656566.9.11.1935. PMID 18627331
- [Background] Roberts AC, Porter KE. Cellular and molecular mechanisms of endothelial dysfunction in diabetes. Diab Vasc Dis Res. 2013 Nov;10(6):472-82. doi: 10.1177/1479164113500680. Epub 2013 Sep 3. PMID 24002671
- [Background] Pacher P, Beckman JS, Liaudet L. Nitric oxide and peroxynitrite in health and disease. Physiol Rev. 2007 Jan;87(1):315-424. doi: 10.1152/physrev.00029.2006. PMID 17237348